CLINICAL TRIAL: NCT01011998
Title: A Phase II Study of Imatinib and Valproic Acid in Patients With CML
Brief Title: A Study of Imatinib and Valproic Acid in Patients With Chronic Myelogenous Leukemia (CML)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn due to lack of accrual per Center DSMP, with PI concurrence
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 0901
Record Dates: First submitted 2009-11-05; First posted 2009-11-11 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-07

CONDITIONS: Chronic Myelogenous Leukemia
Keywords: CML; Chronic Myelogenous leukemia; INST 0901; imatinib; valproic acid; Gleevec
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Gleevec (imatinib), valproic acid — Valproic acid: 250 mg three times per day and then adjusted according to attain a therapeutic level.
  Gleevec will be continued at the dose the patient was taking at the time of entry onto the study.
  Other Names: Valproic acid; Imatinib; Gleevec

SUMMARY:
The aim of this study is to test the effect of the combination of valproate in combination with imatinib with an aim of achieving a maximal molecular response as the primary goal.

DETAILED DESCRIPTION:
The aim of this study is to test the effect of the combination of valproate in combination with imatinib with an aim of achieving a maximal molecular response as the primary goal. Briefly, patients with CML who are taking imatinib and have been found to have a plateau in their level of the bcr-abl transcript will be eligible to participate in the study. Valproate will then be added to the imatinib, and subsequent bcr-abl transcripts will be monitored to see if the addition of valproate produced a further reduction. Patients will be monitored for efficacy and toxicity.

ELIGIBILITY:
Inclusion Criteria:

* All patients, 18 years of age or older, with a diagnosis of CML.
* Patients must have a life expectancy of at least 12 weeks.
* Patients must have an ECOG performance status of 0-2.
* Patients must sign an informed consent.
* Patients should have adequate hepatic function with a total bilirubin < 2 mg/dl and SGOT or SGPT < two times the upper limit of normal, and adequate renal function as defined by a serum creatinine < 1.5 x upper limit of normal.
* Patients with CML in chronic phase on imatinib as first line therapy who fulfill the following criteria:
* The patient has at least two tests for quantitative reverse transcriptase polymerase chain reaction (RT-PCR) for bcr-abl (peripheral blood or bone marrow aspirate). The results of these tests should demonstrate a relative plateau in the effect of imatinib on the detected level of the transcript (i.e. there should less than a ½ log difference between the last two values). Note: Patients will be eligible if the more recent study is greater than the previous study by any value.
* The last two quantitative RT-PCR studies should be at least 3 months apart.
* The patient should have received at least 9 months of imatinib since the diagnosis of CML.
* The patient is tolerating imatinib without any grade 3 or greater toxicity.

Exclusion Criteria:

* Pregnant women or nursing mothers are not eligible for this trial. Patients of child bearing potential must use adequate contraception.
* Patients may receive no other concurrent chemotherapy or radiation therapy during this trial.
* Patients with severe medical problems such as uncontrolled diabetes mellitus or cardiovascular disease or active infections are not eligible for this trial.
* Patients who have a hypersensitivity to valproic acid, derivatives, or any component of the formulation. Patients with hepatic disease or significant impairment, or urea cycle disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
To measure the effect of the combination of valproate in combination with imatinib with an aim of achieving a maximal molecular response as the primary goal. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ian Rabinowitz, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Cancer Center, Albuquerque, New Mexico, United States